CLINICAL TRIAL: NCT06658158
Title: Effects of Cognitive Correction and Stimulus Control in Chronic Insomnia Patients With Sleep Cognitive Distortions and Maladaptive Sleep Patterns
Brief Title: Effects of Cognitive Correction and Stimulus Control in Chronic Insomnia Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CC+SC-insomnia
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Chronic Insomnia
Keywords: chronic insomnia; cognitive correction; stimulus control; sleep hygiene education
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive correction and stimulus control (Experimental)
  Interventions: Behavioral: Cognitive correction and stimulus control
- Sleep hygiene education (Active Comparator)
  Interventions: Behavioral: Sleep hygiene education

INTERVENTIONS:
Behavioral: Cognitive correction and stimulus control — Cognitive correction:
  a) correcting unrealistic sleep expectations; b) maintaining a natural sleep onset; c) avoiding worry about losing control oversleep; d) not associating nocturnal dreaming with adverse daytime consequences; e) avoiding feelings of frustration due to one night of poor sleep; f) developing tolerance to the impact of insomnia and avoiding compensatory behaviors.
  Stimulus control:
  1. Minimize wakefulness during time in bed and establish a positive association between sleepiness and the bed.
  2. Use the bed only for sleep and sexual activities.
  3. Go to bed only when feeling sleepy at night or at the designated sleep time.
  4. If unable to fall asleep within approximately 20 minutes of being in bed, leave the bedroom, engage in relaxing activities, and return to bed when feeling sleepy. Repeat this process if unable to fall asleep within approximately 20 minutes.
  5. Wake up at the same time every morning, including weekends.
  Arms: Cognitive correction and stimulus control
Behavioral: Sleep hygiene education — 1. Sleep until feeling refreshed the next day.
  2. Maintain regular exercise and eating habits, avoiding going to bed on an empty stomach.
  3. Ensure a comfortable bedroom environment with suitable nighttime temperature, free from light and noise disturbances.
  4. Avoid excessive consumption of beverages, alcohol, and smoking at night, and reduce caffeine intake.
  5. Avoid bringing problems to bed and refrain from attempting to sleep.
  6. Place the alarm clock under the bed or move it away from sight.
  7. Avoid daytime napping.
  Arms: Sleep hygiene education

SUMMARY:
This study aims to validate the effect of cognitive correction and stimulus control on correcting sleep cognitive distortions and improving maladaptive sleep behaviors.

DETAILED DESCRIPTION:
Cognitive correction aims to identify and change patients' erroneous beliefs and attitudes about sleep, which may include exaggerated sleep needs, excessive worry about the consequences of insomnia, and unrealistic expectations about bedtime. Stimulus control, on the other hand, focuses on modifying patients' behaviors in bed, linking the bed with a rapid onset of sleep, and reducing the negative association between the bed and insomnia.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the diagnostic criteria for insomnia disorder according to DSM-5;
2. PSQI total score > 5;
3. Age ≥ 18 years, with at least a junior high school education;
4. Sleep cognitive distortions assessed using the DBAS-16;
5. "Maladaptive Sleep Behavior Questionnaire - 8 items" used to assess "maladaptive sleep behaviors";
6. Willing to participate in the study and sign an informed consent form.

Exclusion Criteria:

1. Presence of severe physical illness or serious mental disorders, or at risk for suicide;
2. Clinically diagnosed or suspected sleep-related breathing disorders, restless legs syndrome, and circadian rhythm sleep-wake disorders; shift workers;
3. Pregnant or lactating women;
4. Currently undergoing any form of psychological therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The change of Pittsburgh Sleep Quality Index (PSQI) total scores from baseline to 6 weeks. | Baseline, 6 weeks
  The PSQI consists of 7 factors ranging from 0 to 3 points, and the total score ranges from 0 to 21 with higher scores indicating poorer quality.

SECONDARY OUTCOMES:
The change of PSQI total scores from baseline to 3 months, 6 months, and 12 months. | Baseline, 3 months, 6 months, 12 months
  The PSQI consists of 7 factors ranging from 0 to 3 points, and the total score ranges from 0 to 21 with higher scores indicating poorer quality.
The change of Insomnia severity index (ISI) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The ISI reporting insomnia symptoms severity consists of 7-items on a 5-point Likert scale, and the total score ranges from 0 to 28 with higher scores indicating more severe insomnia.
The change of sleep efficiency from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  Sleep efficiency is assessed with the Carney (2012) consensus sleep diary. This is measured in percentage (higher scores indicating better sleep efficiency).
The change of Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The DBAS assessing sleep related cognitions in 16 items rated on a 10-point Likert scale, and the total score ranges from 0 to 160 with higher scores indicating more intensive dysfunctional beliefs.
The change of Snaith-Hamilton Pleasure Scale (SHAPS) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The SHAPS assessing anhedonia consists of 14 items, and the total score ranges from 14 to 56 with higher scores indicating more serious the anhedonia.
The change of Short Form 36 (SF-36) total scores from baseline to 6 weeks, 3 months, 6 months, 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months.
  The SF-36 quantifying the quality of life in relation to health status consists of 36-items with eight areas covering physical functioning, role limitations brought on by physical issues, bodily pain, general health perceptions, vitality, social functioning, role limitations brought on by emotional issues, and perceived mental health. The total score ranges from 0-100 (the worst possible to the most possible).
The change of Patient Health Questionnaire-4 (PHQ-4) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The PHQ-4 comprises a 2-item depression scale and a 2-item anxiety scale. Each instrument can reach values from 0-6. Higher Scores are indicating higher distress.
The change of Beck Depression Inventory (BDI) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The BDI assessing the existence and severity of symptoms of depression consists of 21 items, and the total score ranges from 0 to 63 with higher scores indicating more severe depressive symptoms.
The change of Beck Anxiety Inventory (BAI) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The BAI assessing the existence and severity of symptoms of anxiety consists of 21 items, and the total score ranges from 0 to 63 with higher scores indicating more severe anxiety.
The change of Patient Health Questionnaire-15 (PHQ-15) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The PHQ-15 measuring somatic distress consists of 15 items, and the total score ranges from 0 to 30 with higher scores indicating more severe somatic distress.
The change of 5-item Perceived Deficits Questionnaire-Depression (PDQ-D-5) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The PDQ-D-5 assessing perceived cognitive deficits from the patient's perspective consists of 5 items, and the total score ranges from 0 to 20 with higher scores indicating greater perceived deficit.
The change of Life Events Scale (LES) total scores from baseline to 3 months, 6 months, 12 months, 18 months, and 24 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The LES assessing the perceived stress and number of stressful life events experienced consists of 48 items which are classified into three dimensions: family life events (28 items), work and study events (13 items), and social events (7 items) with higher scores in LES perceived greater stressfulness.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No